CLINICAL TRIAL: NCT03909854
Title: Pragmatic Investigation of Volume Targeted Ventilation-1 (PIVOT-1)
Brief Title: Pragmatic Investigation of Volume Targeted Ventilation-1
Acronym: PIVOT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00055128
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Failure; Acute Respiratory Distress Syndrome (ARDS); Ventilator Lung
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: Before-and-after trial design of adaptive pressure control and assist volume control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive Pressure Control (Active Comparator): The Adaptive Pressure Control arm is the baseline mode/protocol for medical intensive care unit mechanical ventilation
  Interventions: Procedure: mode of mechanical ventilation
- Assist Volume Control (Active Comparator): The assist volume control arm is the new protocol that will be implemented and tested for feasibility
  Interventions: Procedure: mode of mechanical ventilation

INTERVENTIONS:
Procedure: mode of mechanical ventilation — Adaptive Pressure Control mechanical ventilation is a dual controlled mode that is designed to auto-control flow and minimize inspiratory pressure while delivering a provider-determined tidal volume. Assist Volume Control mechanical ventilation is a mode in which the respiratory care provider determines patient tidal volume and flow.

SUMMARY:
This proposal will test the feasibility of implementing an assist volume control ventilation protocol in patients receiving mechanical ventilation in the medical intensive care unit. The trial will consist of a before-and-after trial design of block assignment to either adaptive pressure control (baseline) or assist volume control .

This is a feasibility study looking at the management of patients in the ventilator.

DETAILED DESCRIPTION:
Over the course of 6 weeks, a before-and-after trial design of adaptive pressure control and assist volume control will be conducted.

Pre-trial planning phase: study protocols will be reviewed with key stakeholders (respiratory therapy providers and medical teams)

Weeks 1-2: data will be collected on our current adaptive pressure control ventilator protocol.

Week 3: The investigators will implement an assist volume control protocol. . Patients already on mechanical ventilation will be converted to assist volume control; however, these patients will not be included in the primary analysis.In accordance with the Consolidated Framework For Implementation Research (CFIR) approach, after 1 week of assist volume control the investigators will engage in quantitative and qualitative feedback with care providers to identify facilitators and barriers of assist volume control implementation.

Week 4-6: If the investigators identify substantial barriers, the investigators will pause and alter the protocol. If not, the investigators will continue assist volume control for an additional 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Acute Respiratory Failure requiring mechanical ventilation medical intensive care unit admission

Exclusion Criteria:

chronic mechanical ventilation clinician use of non-volume-targeted ventilation as initial mode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving Assist Volume Control | 1 hour
  The primary outcome for the PIVOT-1 pilot is feasibility of Assist Volume Control implementation. We define feasibility in this study as 80% of patients receiving Assist Volume Control within 1 hour of initiation of intensive care unit mechanical ventilation

SECONDARY OUTCOMES:
assist volume control duration | 24 hours
  A secondary feasibility outcome will be >70% of ventilated time on Assist Volume Control during the first 24 hours of mechanical ventilation.
Percentage of mode crossover | 2 weeks
  A secondary feasibility outcome will include <10% crossover to the alternative mode
exhaled tidal volume | 2 weeks
  exhaled tidal volume will be compared between modes using data extracted from the critical care data capsule.
Number of ventilator free days | 28 days
  vent free days will be compared between the modes using data from the critical care data analytics platform
intensive care length of stay | 28 days
  intensive care unit length of stay will be compared between the modes using data from the critical care data analytics platform

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Gibbs, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Esteban A, Frutos-Vivar F, Muriel A, Ferguson ND, Penuelas O, Abraira V, Raymondos K, Rios F, Nin N, Apezteguia C, Violi DA, Thille AW, Brochard L, Gonzalez M, Villagomez AJ, Hurtado J, Davies AR, Du B, Maggiore SM, Pelosi P, Soto L, Tomicic V, D'Empaire G, Matamis D, Abroug F, Moreno RP, Soares MA, Arabi Y, Sandi F, Jibaja M, Amin P, Koh Y, Kuiper MA, Bulow HH, Zeggwagh AA, Anzueto A. Evolution of mortality over time in patients receiving mechanical ventilation. Am J Respir Crit Care Med. 2013 Jul 15;188(2):220-30. doi: 10.1164/rccm.201212-2169OC. PMID 23631814
- [Background] Mireles-Cabodevila E, Chatburn RL. Work of breathing in adaptive pressure control continuous mandatory ventilation. Respir Care. 2009 Nov;54(11):1467-72. PMID 19863830
- [Background] Wunsch H, Wagner J, Herlim M, Chong DH, Kramer AA, Halpern SD. ICU occupancy and mechanical ventilator use in the United States. Crit Care Med. 2013 Dec;41(12):2712-9. doi: 10.1097/CCM.0b013e318298a139. PMID 23963122
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Shah FA, Girard TD, Yende S. Limiting sedation for patients with acute respiratory distress syndrome - time to wake up. Curr Opin Crit Care. 2017 Feb;23(1):45-51. doi: 10.1097/MCC.0000000000000382. PMID 27898439
- [Background] Branson RD, Chatburn RL. Controversies in the critical care setting. Should adaptive pressure control modes be utilized for virtually all patients receiving mechanical ventilation? Respir Care. 2007 Apr;52(4):478-85; discussion 485-8. PMID 17417981
- [Background] Figueroa-Casas JB, Montoya R. Effect of Tidal Volume Size and Its Delivery Mode on Patient-Ventilator Dyssynchrony. Ann Am Thorac Soc. 2016 Dec;13(12):2207-2214. doi: 10.1513/AnnalsATS.201605-362OC. PMID 27598383
- [Background] Kallet RH, Campbell AR, Dicker RA, Katz JA, Mackersie RC. Work of breathing during lung-protective ventilation in patients with acute lung injury and acute respiratory distress syndrome: a comparison between volume and pressure-regulated breathing modes. Respir Care. 2005 Dec;50(12):1623-31. PMID 16318643
- [Background] Yoshida T, Fujino Y, Amato MB, Kavanagh BP. Fifty Years of Research in ARDS. Spontaneous Breathing during Mechanical Ventilation. Risks, Mechanisms, and Management. Am J Respir Crit Care Med. 2017 Apr 15;195(8):985-992. doi: 10.1164/rccm.201604-0748CP. PMID 27786562
- [Background] Writing Group for the PReVENT Investigators; Simonis FD, Serpa Neto A, Binnekade JM, Braber A, Bruin KCM, Determann RM, Goekoop GJ, Heidt J, Horn J, Innemee G, de Jonge E, Juffermans NP, Spronk PE, Steuten LM, Tuinman PR, de Wilde RBP, Vriends M, Gama de Abreu M, Pelosi P, Schultz MJ. Effect of a Low vs Intermediate Tidal Volume Strategy on Ventilator-Free Days in Intensive Care Unit Patients Without ARDS: A Randomized Clinical Trial. JAMA. 2018 Nov 13;320(18):1872-1880. doi: 10.1001/jama.2018.14280. PMID 30357256
- [Background] Serpa Neto A, Simonis FD, Barbas CS, Biehl M, Determann RM, Elmer J, Friedman G, Gajic O, Goldstein JN, Horn J, Juffermans NP, Linko R, de Oliveira RP, Sundar S, Talmor D, Wolthuis EK, de Abreu MG, Pelosi P, Schultz MJ. Association between tidal volume size, duration of ventilation, and sedation needs in patients without acute respiratory distress syndrome: an individual patient data meta-analysis. Intensive Care Med. 2014 Jul;40(7):950-7. doi: 10.1007/s00134-014-3318-4. Epub 2014 May 9. PMID 24811940
- [Background] Semler MW, Self WH, Wanderer JP, Ehrenfeld JM, Wang L, Byrne DW, Stollings JL, Kumar AB, Hughes CG, Hernandez A, Guillamondegui OD, May AK, Weavind L, Casey JD, Siew ED, Shaw AD, Bernard GR, Rice TW; SMART Investigators and the Pragmatic Critical Care Research Group. Balanced Crystalloids versus Saline in Critically Ill Adults. N Engl J Med. 2018 Mar 1;378(9):829-839. doi: 10.1056/NEJMoa1711584. Epub 2018 Feb 27. PMID 29485925
- [Background] Casey JD, Janz DR, Russell DW, Vonderhaar DJ, Joffe AM, Dischert KM, Brown RM, Zouk AN, Gulati S, Heideman BE, Lester MG, Toporek AH, Bentov I, Self WH, Rice TW, Semler MW; PreVent Investigators and the Pragmatic Critical Care Research Group. Bag-Mask Ventilation during Tracheal Intubation of Critically Ill Adults. N Engl J Med. 2019 Feb 28;380(9):811-821. doi: 10.1056/NEJMoa1812405. Epub 2019 Feb 18. PMID 30779528
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Zuidgeest MGP, Goetz I, Groenwold RHH, Irving E, van Thiel GJMW, Grobbee DE; GetReal Work Package 3. Series: Pragmatic trials and real world evidence: Paper 1. Introduction. J Clin Epidemiol. 2017 Aug;88:7-13. doi: 10.1016/j.jclinepi.2016.12.023. Epub 2017 May 24. PMID 28549929
- [Background] Meinecke AK, Welsing P, Kafatos G, Burke D, Trelle S, Kubin M, Nachbaur G, Egger M, Zuidgeest M; work package 3 of the GetReal consortium. Series: Pragmatic trials and real world evidence: Paper 8. Data collection and management. J Clin Epidemiol. 2017 Nov;91:13-22. doi: 10.1016/j.jclinepi.2017.07.003. Epub 2017 Jul 14. PMID 28716504
- [Background] Sjoding MW, Gong MN, Haas CF, Iwashyna TJ. Evaluating Delivery of Low Tidal Volume Ventilation in Six ICUs Using Electronic Health Record Data. Crit Care Med. 2019 Jan;47(1):56-61. doi: 10.1097/CCM.0000000000003469. PMID 30308549

DOCUMENTS (1):
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03909854/ICF_000.pdf